CLINICAL TRIAL: NCT06256796
Title: Evaluation of Effectiveness of Fresh Frozen Plasma Transfusion as a Novel Adjuvant Treatment in Acute Organophosphate Poisoned Patients. A Randomized Clinical Trial in Poison Control Center Ain Shams University Hospital.
Brief Title: Fresh Frozen Plasma Transfusion in Acute Organophosphate Poisoning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: plasma in OP poisoning
Record Dates: First submitted 2024-01-22; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-01

CONDITIONS: Organophosphorus Poisoning
MeSH Terms: conditions — Organophosphate Poisoning

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- moderate group controlled patients (No Intervention)
- moderate group study patients (Experimental)
  Interventions: Other: fresh frozen plasma
- sever controlled group (No Intervention)
- sever study group (Experimental)
  Interventions: Other: fresh frozen plasma

INTERVENTIONS:
Other: fresh frozen plasma — repeated doses of fresh plasma over 3 days in organophosphate poisoned patients
  Arms: moderate group study patients; sever study group

SUMMARY:
this study clinical trial to assess the role of fresh frozen plasma as a novel available and easy to be applied rather than conventional therapy on organophosphate poisoned patients and prediction of it is prognosis on selected patients and it is effect on outcome .

DETAILED DESCRIPTION:
a prospective randomized clinical trail study . this study will be conducted in poison control center Ain shas university hospital -Egypt . all adult patients of both sexes admitted , in Poison Control Center of Ain Shams University Hospitals (PCC-ASUH) with diagnosis of moderate and severe degree of organophosphate poisoning will be included in this study.

The severity of patients under the study will be assessed at the time of presentation using the PeradeniyaOrganophosphorus Poisoning (POP) scale The severity will be graded as mild(0-3), moderate (4-7), and sever (8- 11).

The included patients in this study will be randomly divided into two groups as follow:

Group A: Patients who will be treated according to traditional management protocol of OPC toxicity in the form of: supportive measures, decontamination and antidotal therapy (atropine &Oximes) as follow:

* Supportive measures and patients resuscitation.
* Decontamination: patients presenting within 4hr of OP ingestion will be subjected to gastric lavage and all patients with oral exposure will be given a single (30 mg) dose of activated charcoal. Any contaminated material will be discarded and dermal contamination will be carried out using soap and water,if necessary.
* Antidotal therapy: Atropine(each ampoule contains 1mg of atropine per ml) will be given as bolus doses of 2-5 mg IV and repeated every10-15 min until dryness of chest secretions, and then atropine injections maintenance doses will be given intermittently to patients as needed .Toxogonin (each ampoule contains 250mg of obidoxime chloride in 1 ml, produced by Merck, Darmstadt, Germany)will be administered as a loading dose of 250 mg, and will be repeated every 8 hrs until at least 12hrs after atropine no longer required.

This group of patients will be divided in to :

GroupA1 will include moderate degree of acute OP poisoned patients (POP scale 4-7) Group A2 will include severe degree of acute OP poisoned patients (POP scale 8-11)

Group B: Patients who will be treated with conventional therapy of OPC toxicity in the form of: supportive measures, decontamination and antidotal therapy (atropine &Oximes) in addition to fresh frozen plasma (FFP).

FFP will be given after one hour of hospitalization (time needed to prepare FFP to the patients and to finish emergency management) in dose of 20ml\kg given as follows:

* 4 units first day
* 3 units on second day 2 units on third day (

ELIGIBILITY:
Inclusion Criteria:

-moderate and severe degree of organophosphate poisoning will be included in this study.

Exclusion Criteria:

* patients below 18 years or above 60 years.
* Patients with history of diabetes, cardiac disease, respiratory, renal disease and hepatic disease.
* Pregnant female
* Patients suspected of having mixed or unknown exposure
* Patients with coagulation disorders.
* Patients with hyper sensitivity to FFP or plasma derived products, as these cases are contraindicated to take fresh frozen plasma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
mortality rate | 3 monthes
  fresh frozen plasma decrease the mortality rate among organophosphate poisoned patients

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of medicine Ain Shams University, Cairo, Egypt

REFERENCES:
- [Background] Dayananda VP, Bhaskara B, Pateel GN. A study of effectiveness of fresh frozen plasma in organophosphorous compound poisoning in reducing length of Intensive Care Unit stay and in reducing need for tracheostomy. Anesth Essays Res. 2016 May-Aug;10(2):268-72. doi: 10.4103/0259-1162.171455. PMID 27212759